CLINICAL TRIAL: NCT00531037
Title: Natural Evolution of AV Conduction Disorders in Patients Implanted With Cardiac Pacemakers
Acronym: NATURE
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: Nature - RGST01; RGST01
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Patients Implanted With a Pacemaker
Keywords: AV block, SND, BTS, AAIsafeR, SafeR, PM implanted
MeSH Terms: conditions — Atrioventricular Block; Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational study to assess AV block incidence and their evolution according to paroxysmal atrial arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Sinus Node Disease
* Brady-Tachy Syndrome
* Suspected or documented paroxysmal AVB

Exclusion Criteria:

* Permanent high degree AVB
* Contra indication to the SafeR pacing mode
* PR higher than 350 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient primo-implanted with a pacemaker (Symphony ™ DR2550, Symphony ™ D 2450, Reply DR, Reply D or any similar or higher range) device less than three months ago, programmed in SafeR mode.
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
High degree AV blocks | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: DEHARO Jean Claude, MD, Principal Investigator — CHU la Timone - Marseille
Locations (129):
- United States (7):
  - Baptist Princeton Birmingham, Birmingham, Alabama
  - Tennessee Valley Sheffield, Sheffield, Alabama
  - Cardiovascular Assoc. Of Mesa, Mesa, Arizona
  - O'Connor Hospital San Jose, San Jose, California
  - Piedmont hospital, Piedmont, Georgia
  - University of Mississippi Medical Center, Mississippi City, Mississippi
  - St. Francis Hospital Tulsa, Tulsa, Oklahoma
- Belgium (3):
  - Az St- Blasius, Dendermonde
  - Ch de Huy, Huy
  - Heilig Hart Ziekenhuis MOL, Mol
- Canada (2):
  - Hospital Hamilton, Hamilton
  - Niagara Health System, Niagara
- Denmark (2):
  - Bispebjerg Hospital, Bispebjerg
  - HELLERUP, Gentofte Hospital
- France (80):
  - Clinique Esquirol, Agen
  - CH Albi, Albi
  - Clinique Claude Bernard, Albi
  - CH ALES, Alès
  - Clinique Bonnefond, Alès
  - Cabinet Prive, Annecy
  - Clinique Aressy, Aressy
  - CH AUCH, Auch
  - Clinique Paulmy, Bayonne
  - Ch Beauvais, Beauvais
  - Clinique St Vincent, Besançon
  - Ch Beziers, Béziers
  - Clinique Aguilera, Biarritz
  - Chu Pessac, Bordeaux
  - Clinique Des Pins Francs, Bordeaux
  - Ch Boulogne, Boulogne-sur-Mer
  - Chu Brest, Brest
  - CH BRIVE, Brivé
  - Ch Calais, Calais
  - Clinique Des 2 Caps, Calais
  - Ch Carcassonne, Carcassonne
  - Chu Ceret, Ceret
  - Ch Chaumont, Chaumont
  - Ch Chalons, Châlons-en-Champagne
  - Clinique Bon Secours, Châtellerault
  - Ch Cherbourg, Cherbourg
  - Ch Colmar, Colmar
  - Cabinet Cardiologie Creutzwald, Creutzwald
  - Polyclinique Du Parc, Croix
  - CH DINAN, Dinan
  - CH DOLE, Dole
  - CH DOUAI, Douai
  - Ch Douarnenez, Douarnenez
  - Polyclinique Notre Dame, Draguignan
  - Hôpital Emile Roux, Eaubonne
  - Centre Cardiologique D'Evecquemont, Évecquemont
  - Hôpital D'Evreux, Évreux
  - Ch Firminy, Firminy
  - Ch Forbach, Forbach
  - Ch Freyming, Freyming-Merlebach
  - CH GAP, Gap
  - Ch Lannion, Lannion
  - Cmc Parly Ii, Le Chesnay
  - Ch Le Havre, Le Havre
  - Chu Le Havre, Le Havre
  - Centre Medico Chirurgical de L'Europe, Le Port-Marly
  - Hôpital Cardiologique, Lyon
  - Chu La Timone, Marseille
  - Hôpital Nord, Marseille
  - Chg Martigues, Martigues
  - Institut Hospitalier Jacques Cartier, Massy
  - Hôpital Ste Blandine, Metz
  - Clinique Pont Chaume, Montauban
  - Hôpital Le Raincy Monfermeil, Montfermeil
  - Chu Montpellier, Montpellier
  - Clinique Plein Ciel, Mougins
  - Ch Moulins, Moulins
  - Clinique Du Diaconnat, Mulhouse
  - Centre Chirurgical Ambroise Pare, Neuilly-sur-Seine
  - Ch Nevers, Nevers
  - Clinique Des Fleurs, Ollioules
  - Ch Orange, Orange
  - Clinique Bizet, Paris
  - Clinique Parc Monceau, Paris
  - Hôpital Val de Grâce, Paris
  - CHU PAU, Pau
  - Ch Perpignan, Perpignan
  - Chu Poitiers, Poitiers
  - Hôpital Prive Claude Galien, Quincy-sous-Sénart
  - Clinique Pasteur, Ris-Orangis
  - CH RODEZ, Rodez
  - Clinique St Hilaire Rouen, Rouen
  - Polyclinique de Montier La Celle, Saint-André-les-Vergers
  - Centre Cardiologique Du Nord, Saint-Denis
  - Clinique Notre Dame, Saint-Dié
  - Hôpital Prive Nord Parisien, Sarcelles
  - Ch St Malo, St-Malo
  - Cmc Ste Feyre, STE Feyre
  - Clinique St Gatien, Tours
  - Clinique Vauban, Valenciennes
- Germany (5):
  - Erzgebirgsklinikum ANNABERG, Annaberg
  - Schade Stolz Rötech, Berlin
  - Klinikum Bogenhausen, Bogenhausen
  - Klinikum Dresden, Dresden
  - PRAXIS Dr Subin und Lutter, Hamburg
- Italy (3):
  - Hospital Montebelluna, Montebelluna
  - Hospital Negrar, Negrar
  - Casa di Cura Pederzoli, Peschiera del Garda
- Japan (11):
  - Kanagawa Cardiov. and Respiratory Center, Kanagawa
  - Kokura Memorial Hospital, Kokura
  - Konan St Hill Hospital, Kōnan
  - Yokosuka Kyosai General Hospital, Kyosai
  - Mie University Hospital, Mie
  - Nara Hospital, Kinki University School of Medicine, Nara
  - Ogikubo Hospital, Ogikubo
  - Saiseikai Noe Hospital, Saiseikai NOE
  - Tokio Metropolitan Geriatric Hospital, Tokyo
  - Tokai University School of Medicine, Tōkai
  - Yokohama City University Hospital, Yokohama
- Portugal (8):
  - Hospital de Santa Cruz, Carnaxide, Lisbon District
  - Hospital Garcia Orta, Almada
  - Hospital Central Faro, Faro
  - Hospital Egas Moniz, Lisbon
  - Hospital Santa Maria, Lisbon
  - Hospital Santa Marta, Lisbon
  - Hospital São Francisco Xavier, Lisbon
  - Hospital Distrital de Santarém, Santarém
- Seoul National University Hospital, Seoul, South Korea
- Spain (7):
  - Hospital Marina Alta, Denia
  - Hospital General de Elda, Elda
  - Hospital de Cabuenes, Gijón
  - Hospital Vega Baja, Orihuela
  - Hospital Arnau de Vilanova, Valencia
  - Hospital La Fe, Valencia
  - Meixoeiro, Vigo